CLINICAL TRIAL: NCT01660399
Title: Boanmycin Hydrochloride for Injection in Combination With Docetaxel for Patients With Advanced Lung Squamous Cell Carcinoma as Salvage Chemotherapy: a Prospective, Randomized, Parallel and Controlled Clinical Trial
Brief Title: Clinical Trial of Boanmycin Hydrochloride With Docetaxel for Patients With Lung Squamous Cell Cancer as Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIH-CHP-201205001
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-08

CONDITIONS: Squamous Cell Lung Cancer
Keywords: salvage chemotherapy; advanced squamous cell lung cancer; Boanmycin
MeSH Terms: interventions — bleomycin A6; Injections; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel/Boanmycin (Experimental): Docetaxel 75mg/m2, intravenous infusion, day 1; Boanmycin 5-6 mg/m2 + DXM 5mg IVD or IM, day 3,5,10,12, 21days a cycle.
  Interventions: Drug: Boanmycin; Drug: Docetaxel
- Docetaxel (Placebo Comparator): Docetaxel 75mg/m2, intravenous infusion, day 1, 21days a cycle.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Boanmycin — Boanmycin 5-6 mg/m2 + DXM 5mg IVD or IM, day 3,5,10,12, 21days a cycle.
  Other Names: Boanmycin Hydrochloride for Injection
  Arms: Docetaxel/Boanmycin
Drug: Docetaxel — Docetaxel 75mg/m2, intravenous infusion, day 1.
  Other Names: Docetaxel for Injection

SUMMARY:
This predictive, randomized, double-blind, multi-center trial is going to evaluate the efficacy and safety of two regimens of boanmycin plus docetaxel versus docetaxel alone as a second line treatment for chemotherapy for stage IIIb-IV or postoperative recurrent squamous cell lung cancer patients.

DETAILED DESCRIPTION:
At present, there is no reliable second line treatment except chemotherapy for squamous cell carcinoma patients, the current chemotherapy regimen, including docetaxel as a single agent which is known as the gold standard, the weekly using of docetaxel and the combination of EGFR-TKI has few evidence for high response rates and prolonged survival.On the other hand, the adverse reaction of chemotherapy makes the combined chemotherapy cannot improve therapeutic effects. Boanmycin with special pharmacological basis, as well as the high purity, may not obvious increase in adverse reactions, and probably improve the effect of chemotherapy. At the same time, because of its low lung toxicity, especially in the combined use of corticosteroids, and in the background of the poor survival of advanced squamous cell lung cancer patients, the chemotherapy regimen of boanmycin plus docetaxel needs to be investigated.

This predictive, randomized, double-blind, multi-center trial is going to evaluate the efficacy and safety of two regimens of boanmycin plus docetaxel versus docetaxel alone as a second line treatment for chemotherapy for stage IIIb-IV or postoperative recurrent squamous cell lung cancer patients.

According to the test center, gender, disease staging (stage IIIB, IV/recurrence) and pathologic types, patients with squamous cell lung cancer were stratified and then randomly assigned to one of two groups. In the first group, 75 mg of docetaxel per square meter of body-surface area, administered on day 1, followed by 5~6 mg boanmycin of per square meter and 5mg dexamethasone on days 3,5,10 and 12, the cycle was repeated every 21days. The second group received the reference treatment: docetaxel at a dose of 75 mg per square meter was administered on on day 1 of a three-week cycle. The efficacy was evaluated using RESIST standard after every 2 cycles of the treatment, the regimen will continue until the disease progression or the appearance of not tolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytology confirmed III，IV or after operation recurrent squamous cell lung cancer;
* disease progressed after first-line chemotherapy and not suitable for EGFR-TKI;
* no radiotherapy for metastases outside the lung 4 weeks before;
* the lesions are measurable in CT images and are measured follow criteria RECIST 1.1 2 weeks before randomization;
* ECOG scale 0-1, expected survival>3 month;
* white blood count ≥ 3,500/mm3, absolute neutrophil≥ 1,500/mm3, platelet count ≥ 100,000/mm3, hemoglobin count≥ 90 g/dL；serum bilirubin level ≤ 1.5 of the upper limit of normal(ULN) for the institution, aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase≤ 2.5 ULN, serum creatinine≤ 1.5 ULN;
* with good compliance；

Exclusion Criteria:

* past history of major operation in 4 weeks;
* involved in other clinical trials in 4 weeks;
* past history of central nervous system or relevant disease except for well-controlled CNS metastasis;
* past history of other cancers except for cured non-melanoma skin cancer or cervical cancer;
* concomitant treatment with other anticancer drugs.
* pregnancy, breast feeding or fertility but not taking contraceptive device during the trials;
* radiotherapy for target lesions in lung;
* clear TKI-related mutation in EGFR;
* with severe heart disease, hypertension, diabetes mellitus or active infection.
* past history of allergy to taxanes;
* past history of severe acute or chronic kidney disease;
* active hepatitis b or HIV positive patients;
* cannot tolerate Corticosteroid;
* past history of COPD or other critical basic pulmonary diseases;
* history of severe mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 1.5 years
  DFS was defined as the length of time from the date of randomization to the date of first documentation of relapse of gastric cancer or any other type of cancer or death.

SECONDARY OUTCOMES:
overall survival | 1.5 years
  OS was defined as the length of time from the date of randomization to the date of death of various reasons.

OTHER OUTCOMES:
Adverse Events | 1.5 years
  An Adverse Events is any unfavorable and unintended medical occurrence/sign (including an abnormal laboratory finding), symptom or disease in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
serious adverse event | 1.5 years
  SAE is medically significant or requires intervention to prevent one or other of the outcomes, such as: Fatal (results in death);Life-Threatening Hospitalization; prolong hospitalization; Anomaly/birth defect or Disability/incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Chen, M.D., Principal Investigator — Department of Pulmonary Medical Oncology, Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Pulmonary Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Result] Chemotherapy in non-small cell lung cancer: a meta-analysis using updated data on individual patients from 52 randomised clinical trials. Non-small Cell Lung Cancer Collaborative Group. BMJ. 1995 Oct 7;311(7010):899-909. PMID 7580546
- [Result] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Result] Socinski MA, Schell MJ, Peterman A, Bakri K, Yates S, Gitten R, Unger P, Lee J, Lee JH, Tynan M, Moore M, Kies MS. Phase III trial comparing a defined duration of therapy versus continuous therapy followed by second-line therapy in advanced-stage IIIB/IV non-small-cell lung cancer. J Clin Oncol. 2002 Mar 1;20(5):1335-43. doi: 10.1200/JCO.2002.20.5.1335. PMID 11870177
- [Result] Buter J, Giaccone G. EGFR inhibitors in lung cancer. Oncology (Williston Park). 2005 Nov;19(13):1707-11; discussion 1711-2, 1720-3. PMID 16425523
- [Result] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Result] Eberhard DA, Johnson BE, Amler LC, Goddard AD, Heldens SL, Herbst RS, Ince WL, Janne PA, Januario T, Johnson DH, Klein P, Miller VA, Ostland MA, Ramies DA, Sebisanovic D, Stinson JA, Zhang YR, Seshagiri S, Hillan KJ. Mutations in the epidermal growth factor receptor and in KRAS are predictive and prognostic indicators in patients with non-small-cell lung cancer treated with chemotherapy alone and in combination with erlotinib. J Clin Oncol. 2005 Sep 1;23(25):5900-9. doi: 10.1200/JCO.2005.02.857. Epub 2005 Jul 25. PMID 16043828
- [Result] Pirker R, Pereira JR, Szczesna A, von Pawel J, Krzakowski M, Ramlau R, Vynnychenko I, Park K, Yu CT, Ganul V, Roh JK, Bajetta E, O'Byrne K, de Marinis F, Eberhardt W, Goddemeier T, Emig M, Gatzemeier U; FLEX Study Team. Cetuximab plus chemotherapy in patients with advanced non-small-cell lung cancer (FLEX): an open-label randomised phase III trial. Lancet. 2009 May 2;373(9674):1525-31. doi: 10.1016/S0140-6736(09)60569-9. PMID 19410716
- [Result] Fossella FV, Lee JS, Shin DM, Calayag M, Huber M, Perez-Soler R, Murphy WK, Lippman S, Benner S, Glisson B, et al. Phase II study of docetaxel for advanced or metastatic platinum-refractory non-small-cell lung cancer. J Clin Oncol. 1995 Mar;13(3):645-51. doi: 10.1200/JCO.1995.13.3.645. PMID 7884425
- [Result] Shepherd FA, Dancey J, Ramlau R, Mattson K, Gralla R, O'Rourke M, Levitan N, Gressot L, Vincent M, Burkes R, Coughlin S, Kim Y, Berille J. Prospective randomized trial of docetaxel versus best supportive care in patients with non-small-cell lung cancer previously treated with platinum-based chemotherapy. J Clin Oncol. 2000 May;18(10):2095-103. doi: 10.1200/JCO.2000.18.10.2095. PMID 10811675
- [Result] MA Jinlan, FENG Fengyi, ZHOU Liqiang, SUN Yan.Pharmacokinetics Study and Clinical Evaluation on Boanmycin.China Pharmacy 16(17):1314-1315, 2005.
- [Result] Wang Ping hui, Liu Liping, Hou Yuanshu et al.Phase II Clinical Trial of The New Anticancer Drug-Boanmycin.Chinese Journal of Clinical Oncology 25(9):657-659, 1998.